CLINICAL TRIAL: NCT05279079
Title: International Prospective Evaluation of Novel Biomarkers to Detect and Predict the Severity of Drug- Associated Acute Pancreatitis in Adults
Brief Title: Markers in Acute Pancreatitis-1
Acronym: MAP-1
Status: Active, not recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Innovative Medicines Initiative (Other); TransBioLine Consortium (Unknown); Liverpool University Hospitals NHS Foundation Trust (Other Government); Klinikum der Universität München (Unknown); Hospital Regional de Malaga (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001572
Record Dates: First submitted 2022-02-18; First posted 2022-03-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-07

CONDITIONS: Acute Pancreatitis Drug-Induced
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (10 ml in ethylene diamine tetra-acetic acid, EDTA, 8.5 ml in serum separator tube, SST, 2.5 ml in RNA PAXgene) and urine samples (50 ml collected in Falcon or other tube) will be taken at a single sampling time point from individuals in all groups. These samples will be taken on hospital admission from recruited patients in Groups 1 and 2. Further blood samples (10 ml in EDTA, 8.5 ml in SST and 2.5 ml in RNA PAXgene) will be taken at Day 4 (+/- 1 day) and Day 14 (+/- 2 days) from participants in Groups 1 and 2 from within the United Kingdom.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Group 1: Drug-associated AP: patients aged 18 or more years undergoing drug treatment that has a defined risk of AP prior to and at the onset of AP
  Interventions: Diagnostic Test: Assessment of accuracy of microRNA and pancreatic enzyme markers in blood and/or urine in the detection and/or prediction of severity of drug-associated acute pancreatitis
- Group 2: Other cause AP: patients aged 18 or more years not undergoing drug treatment that has a defined risk of AP prior to and at the onset of AP
  Interventions: Diagnostic Test: Assessment of accuracy of microRNA and pancreatic enzyme markers in blood and/or urine in the detection and/or prediction of severity of drug-associated acute pancreatitis
- Group 3: Chronic pancreatitis: patients aged 18 or more years with symptomatic chronic pancreatitis confirmed by CT or MRI
  Interventions: Diagnostic Test: Assessment of accuracy of microRNA and pancreatic enzyme markers in blood and/or urine in the detection and/or prediction of severity of drug-associated acute pancreatitis
- Group 4: Pancreas cancer: patients aged 18 or more years with biopsy proven pancreas cancer
  Interventions: Diagnostic Test: Assessment of accuracy of microRNA and pancreatic enzyme markers in blood and/or urine in the detection and/or prediction of severity of drug-associated acute pancreatitis
- Group 5: Diabetes mellitus: patients aged 18 or more years with type 1 or type 2 diabetes mellitus in receipt of insulin or oral hypoglycaemics
  Interventions: Diagnostic Test: Assessment of accuracy of microRNA and pancreatic enzyme markers in blood and/or urine in the detection and/or prediction of severity of drug-associated acute pancreatitis
- Group 6: Healthy volunteers
  Interventions: Diagnostic Test: Assessment of accuracy of microRNA and pancreatic enzyme markers in blood and/or urine in the detection and/or prediction of severity of drug-associated acute pancreatitis

INTERVENTIONS:
Diagnostic Test: Assessment of accuracy of microRNA and pancreatic enzyme markers in blood and/or urine in the detection and/or prediction of severity of drug-associated acute pancreatitis — Panel of microRNA and pancreatic enzyme biomarkers

SUMMARY:
Prospective, multi-national, multi-centre observational diagnostic study of novel microRNA and protein biomarkers in peripheral blood and/or urine to detect and predict the severity of drug-associated acute pancreatitis (AP), with comparison of the same biomarkers in patients with acute pancreatitis from other causes, chronic pancreatitis, pancreatic cancer, diabetes mellitus and healthy volunteers.

DETAILED DESCRIPTION:
The MAP-1 study is designed to validate microRNA and/or pancreatic digestive enzyme biomarkers for the detection and severity assessment of drug-associated AP, for application to the assessment of adverse reactions to drugs in development or drugs already developed for other indications. The study will also assess the clinical utility of these biomarkers in AP from other causes, but is not designed to determine whether the biomarkers could be used in place of amylase and/or lipase in the standard clinical diagnosis of AP or to distinguish between the many differential diagnoses of AP. Selection is in progress of the microRNAs and pancreatic digestive enzyme biomarkers to be validated in this study, this selection being made from prospectively biobank samples obtained in a separate observational study that has separate ethical approval.

The pre-selected microRNAs and pancreatic digestive enzymes will be measured in the blood and urine of patients on admission to hospital with drug-associated acute pancreatitis (Group 1, 75 participants in receipt of one or more drugs on a defined list of drugs associated with acute pancreatitis) or other cause acute pancreatitis (Group 2, 250 participants not in receipt of any of the defined drugs). The same biomarkers will also be measured in blood and urine samples from contrast groups of patients with chronic pancreatitis (Group 3, 25 participants), pancreas cancer (Group 4, 25 participants), type I or II diabetes mellitus (Group 5, 25 participants) and healthy volunteers (Group 6, 100 participants). All participants will be at least 18 years old. MicroRNAs will be measured by quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) and pancreatic enzymes by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Drug-associated AP: patients ≥18 years old undergoing drug treatment that has a defined risk of AP prior to and at the onset of AP and admitted to recruiting hospitals with a diagnosis of AP established by two of: (i) typical continuous upper abdominal pain (in this study for up to 2 days in duration prior to admission); (ii) amylase and/or lipase 3 or more times the upper limit of normal; (iii) characteristic findings on abdominal imaging (if undertaken urgently by computerised tomography scan (CT) or magnetic resonance imaging (MRI); and who undergo their first study blood sampling within 24 hours of admission to hospital.
2. Other cause AP: patients ≥18 years old not undergoing drug treatment that has a defined risk of AP and admitted to recruiting hospitals with a diagnosis of AP established by two of: (i) typical continuous upper abdominal pain (in this study for up to 2 days in duration prior to admission); (ii) amylase and/or lipase 3 or more times the upper limit of normal; (iii) characteristic findings on abdominal imaging (if undertaken urgently by CT or MRI) and undergo their first study blood sampling within 24 hours of hospital admission.
3. Chronic pancreatitis: patients with symptomatic chronic pancreatitis and diagnostic abnormalities identified by CT and/or MRI and who undergo study blood sampling as an outpatient.
4. Pancreatic cancer: patients presenting with biopsy-proven or presumed pancreatic cancer and who undergo study blood sampling as an outpatient; in patients with a presumptive diagnosis of pancreatic cancer, blood and urine samples will be analysed after histological confirmation.
5. Diabetes mellitus: adult patients with type 1 or type 2 diabetes mellitus treated with insulin and/or oral anti-hyperglycaemic medication for at least 3 months and ongoing and who undergo study blood sampling as an outpatient.
6. Healthy volunteers: normal, healthy individuals aged ≥18 years old without evidence of systemic disease who have required no hospital intervention within the last year and received no drug treatment within the last 3 months and are severe acute respiratory distress syndrome corona virus 2 (SARS-CoV-2) negative.

Exclusion Criteria:

1. Drug-associated AP: onset of continuous abdominal pain more than 2 days prior to admission to hospital; known previous AP within the last 3 months; known chronic pancreatitis; known pancreatic or hepatobiliary malignancy; previous necrosectomy or pancreatic surgery; known prior type 1 or type 2 diabetes mellitus. Patients will not be excluded if they are undergoing drug treatment that has a defined risk of AP prior to and at the onset of AP and an alternative cause for AP is identified (including after recruitment and blood sampling).
2. Other cause AP: undergoing drug treatment that has a defined risk of AP (such patients should be considered for recruitment into Group 2); onset of continuous abdominal pain more than 2 days prior to admission to hospital; known previous AP within the last 3 months; known chronic pancreatitis; known pancreatic or hepatobiliary malignancy; previous necrosectomy or pancreatic surgery; type 1 or type 2 diabetes mellitus.
3. Chronic pancreatitis: hospital admission with AP within the last three months; known pancreatic or hepatobiliary malignancy; previous necrosectomy or pancreatic surgery; type 1 or type 2 diabetes mellitus.
4. Pancreatic cancer: hospital admission with AP within the last 3 months; known chronic pancreatitis; previous necrosectomy or pancreatic surgery and/or chemotherapy prior to sampling; type 1 or type 2 diabetes mellitus.
5. Diabetes mellitus: hospital admission with AP within the last 3 months; known type 3c diabetes mellitus; known history of acute or chronic pancreatitis; known history of cystic fibrosis, known history of pancreatic or hepatobiliary malignancy; known history of necrosectomy or pancreatic surgery; gestational diabetes mellitus; monogenic diabetes mellitus syndromes; post-transplantation diabetes mellitus; diabetes mellitus attributed to drugs or toxins.
6. Healthy volunteers: abnormal physical examination, abnormal routine haematology, urea, electrolytes and/or liver function tests; evidence of systemic disease; solid or haematological neoplasia within the last 5 years; hospital intervention within last 12 months; scheduled drug treatment within last 3 months and/or as required drug treatment within the last 4 weeks; infection or other sources of acute inflammation within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants aged 18 years or more, comprised of 6 Groups:
  Group 1: Drug-associated AP Group 2: Other cause AP Group 3: Chronic pancreatitis Group 4: Pancreas Cancer Group 5: Diabetes mellitus Grouip 6: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
MicroRNA panel | Day of admission
  Scale of change from normal (healthy volunteer values) of a panel of microRNAs measured in blood and urine samples from patients with mild, moderate or severe drug-associated AP during the first 24 hours of admission, confirming specificity by comparison with results from patients with other pancreatic diseases

SECONDARY OUTCOMES:
Pancreatic enzyme biomarker | Day of admission
  Scale of change from normal (healthy volunteer values) of a selected pancreatic enzyme biomarker in blood and/or urine taken from patients with mild, moderate or severe drug-associated AP during the first 24 hours of admission, confirming specificity by comparison with results from patients with other pancreatic diseases
MicroRNA panel | Days 4 and 14 after admission
  Scale of change of circulating microRNAs measured in blood samples on Day 4 (+/- 1 day) and Day 14 (+/- 2 days) after admission to assess progression of AP
Severity of AP | Within 90 days of admission
  Determination of AP severity will be made according to the Revised Atlanta Classification
Patient reported outcome | Days 4 and 14
  Application of the PAtieNt-rePoRted OutcoMe scale in acute pancreatItis - an international proSpEctive cohort study (PAN-PROMISE) scale
Progress of MAP-1 | Two years
  Progress of recruitment of patients into MAP-1

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sutton, MD FRCS PhD, Principal Investigator — University of Liverpool
Locations (4):
- LMU Klinikum München, Munich, Bavaria, Germany
- Hospital Regional Universitario de Málaga, Málaga, Málaga, Spain
- United Kingdom (2):
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - Aintree University Hospital, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: Undecided